CLINICAL TRIAL: NCT07119619
Title: Evaluation of the Clinical and Radiographic Success of Platelet-Rich Fibrin, Chitosan, and Blood Clot as Scaffolds in Regenerative Endodontic Treatment of Molars
Brief Title: Clinical and Radiographic Outcomes of PRF, Chitosan, and Blood Clot in Regenerative Endodontics of Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Beyza Sandal, Research assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/64; TDH-2023-3161 (Other Grant/Funding Number: Inonu University Scientific Research Projects Unit)
Record Dates: First submitted 2025-06-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Regenerative Endodontics
Keywords: Bllod clot; Chitosan; PRF; Regenerative endodontics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chitosan (Other)
  Interventions: Procedure: Regenerative Endodontic Treatment Using a Chitosan as a Scaffold
- Platelet-rich fibrin (Other)
  Interventions: Procedure: Regenerative Endodontic Treatment Using a Platelet Rich Fibrin as a Scaffold
- Blood clot (Other)
  Interventions: Procedure: Regenerative Endodontic Treatment Using a Blood Clot as a Scaffold

INTERVENTIONS:
Procedure: Regenerative Endodontic Treatment Using a Blood Clot as a Scaffold — During the initial visit, the teeth were anesthetized using inferior alveolar block anesthesia. The endodontic access cavity was then opened. Each canal was irrigated with 2.5% NaOCl and saline. The canals were dried with paper points. Ca(OH)2 was placed in the canals with the objective of achieving an antimicrobial effect. After the application of root canal disinfectant, the opened cavity was sealed with a temporary filling material.The patient has been scheduled for a follow-up appointment within one to four weeks. During the second appointment, local anesthesia was performed using an anesthetic agent that did not contain a vasoconstrictor. The canals were irrigated with 17% EDTA and dried with paper points. Bleeding was induced by instrumentation with a K-type file, at 2 mm past the apical foramen, thus creating a blood clot within the canal. MTA was applied on the scaffold as capping material.
  Arms: Blood clot
Procedure: Regenerative Endodontic Treatment Using a Chitosan as a Scaffold — During the initial visit, the teeth were anesthetized using inferior alveolar block anesthesia. The endodontic access cavity was then opened. Each canal was irrigated with 2.5% NaOCl and saline. The canals were dried with paper points. Ca(OH)2 was placed in the canals with the objective of achieving an antimicrobial effect. After the application of root canal disinfectant, the opened cavity was sealed with a temporary filling material. The patient has been scheduled for a follow-up appointment within one to four weeks.
  During the second appointment, local anesthesia was performed using an anesthetic agent that did not contain a vasoconstrictor. The canals were irrigated with 17% EDTA and dried with paper points.Chitosan in gel form was placed into the root canal space with the help of an injector.MTA was applied on the scaffold as capping material.
  Arms: Chitosan
Procedure: Regenerative Endodontic Treatment Using a Platelet Rich Fibrin as a Scaffold — During the initial visit, the teeth were anesthetized using inferior alveolar block anesthesia. The endodontic access cavity was then opened. Each canal was irrigated with 2.5% NaOCl and saline. The canals were dried with paper points. Ca(OH)2 was placed in the canals with the objective of achieving an antimicrobial effect. After the application of root canal disinfectant, the opened cavity was sealed with a temporary filling material.The patient has been scheduled for a follow-up appointment within one to four weeks. During the second appointment, local anesthesia was performed using an anesthetic agent that did not contain a vasoconstrictor. The canals were irrigated with 17% EDTA and dried with paper points.Ten milliliters of venous blood was collected from the patient and immediately placed in a centrifuge at 3000 rpm for 10 minutes. The prepared PRF was placed in the canal space. MTA was applied on the scaffold as capping material.
  Arms: Platelet-rich fibrin

SUMMARY:
This clinical trial aimed to evaluate the long-term effects of using chitosan, blood clots, and platelet-rich fibrin as scaffolds in regenerative endodontics on tooth development. The trial aimed to answer the following questions:

Does chitosan shorten the duration of treatment for participants? Does chitosan promote root development? Which scaffold is most effective for root development? Which scaffold is more practical and effective to use in pediatric patients? Participants underwent regenerative endodontic treatment and were called to the clinic every six months for symptom assessment. Clinical and radiographic records were kept.

DETAILED DESCRIPTION:
Regenerative endodontic treatments are biologically based procedures designed to physiologically replace damaged tooth structures, including the cells of the pulp-dentin complex. The aim of this treatment is to promote normal root development in immature permanent teeth with necrotic pulp.The primary goal of regenerative endodontics is to stimulate stem cells and encourage their division and proliferation to regenerate damaged tissue. However, a scaffold is essential for the survival of stem cells throughout the regeneration process. A key component of this process is the presence of a scaffold that allows stem cells from the apical papilla to adhere, proliferate, and differentiate. Blood clots and platelet-rich fibrin are frequently used as scaffolds in regenerative endodontics. However, research is ongoing to determine the appropriate scaffold for cases where these are not applicable.Researchers investigated an alternative scaffold for children who could not achieve apical bleeding or allow blood collection from the arm for PRF. Due to its biocompatibility, low cost, and broad-spectrum antibacterial activity, chitosan was included as the third group in this study. The immature necrotic molars to be treated were randomly divided into three groups. Regenerative endodontic treatment was performed using three different scaffolds: blood clot, PRF, and chitosan. The results were evaluated radiographically and clinically.

ELIGIBILITY:
Inclusion Criteria:

Patient Selection Criteria

* Being between the ages of 6-14
* Not having any systemic disease
* Not using any regular medication
* Not having any detected allergies
* The patient must be able to cooperate to the extent that the treatment can be applied healthily
* The patient's guardian must agree to participate in the study

Selection Criteria of Teeth • Restorable necrotic immature first and second permanent mandibular molars with two roots and a root development stage of 3 or 4 according to Cvek's classification

Exclusion Criteria:

• Failure to meet the patient and tooth selection criteria mentioned above

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Radiographic measurements of teeth treated with regenerative endodontic treatment | Baseline and through study completion, an average of 18 months
  Root length and thickness (millimeters)
Radiographic measurements of teeth treated with regenerative endodontic treatment | Baseline and through study completion, an average of 18 months
  Evaluation of root maturation (Cvek score; with a minimum of 1 and a maximum of 5, higher scores mean a better result)

SECONDARY OUTCOMES:
Radiographic measurements of teeth treated with regenerative endodontic treatment | Baseline and through study completion, an average of 18 months
  Periapical healing (Periapical index; with a minimum of 1 and a maximum of 5, lower scores mean a better result)

CONTACTS AND LOCATIONS:
Overall Officials: Beyza Sandal, Study Chair — Derince Oral and Dental Health Center
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cehreli ZC, Isbitiren B, Sara S, Erbas G. Regenerative endodontic treatment (revascularization) of immature necrotic molars medicated with calcium hydroxide: a case series. J Endod. 2011 Sep;37(9):1327-30. doi: 10.1016/j.joen.2011.05.033. Epub 2011 Jul 13. PMID 21846559
- [Background] Ulusoy AT, Turedi I, Cimen M, Cehreli ZC. Evaluation of Blood Clot, Platelet-rich Plasma, Platelet-rich Fibrin, and Platelet Pellet as Scaffolds in Regenerative Endodontic Treatment: A Prospective Randomized Trial. J Endod. 2019 May;45(5):560-566. doi: 10.1016/j.joen.2019.02.002. Epub 2019 Mar 30. PMID 30935618

DOCUMENTS (3):
  • Study Protocol (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT07119619/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT07119619/SAP_001.pdf
  • Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT07119619/ICF_002.pdf